CLINICAL TRIAL: NCT01875276
Title: Evaluating the Need for a New Combination Nasal Spray in the Treatment of Seasonal Rhinitis
Brief Title: Evaluating the Need for New Rhinitis Treatment
Acronym: MEDA
Status: Completed | Type: Observational
Sponsor: Research in Real-Life Ltd (Network)
Collaborators: Meda Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, David Price, Prof., MD, Professor David Price, Research in Real-Life Ltd
Other Study IDs: R04412
Record Dates: First submitted 2013-06-07; First posted 2013-06-11 (Estimated); Last update posted 2013-06-11 (Estimated); Status verified 2013-06

CONDITIONS: Rhinitis
Keywords: Rhinitis; Antihistamine; Nasal Steroid Therapy
MeSH Terms: conditions — Rhinitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Persistent Patients: Defined as those with ≥1 treatment for allergic rhinitis in the six months preceding the IPD (defined as the first script of the hay fever season - May to August)
- Seasonal Rhinitis: No treatment for allergic rhinitis in the six months preceding the IPD

SUMMARY:
The proposed study will evaluate the unmet therapy need in seasonal rhinitis by aiming to answer the following research questions

1. What is the first prescription of the hay-fever season and how many of these patients are on some form of combination therapy?
2. To what extent does initial therapy not meet clinical need (as measured by need for additional medical intervention in terms of consultations and changes in therapy)?
3. Does treatment for allergic rhinitis differ for asthma Vs non-asthma and seasonal Vs perennial patients?

DETAILED DESCRIPTION:
Allergic rhinitis is a chronic respiratory disease with a major impact on quality of life. In a study looking at the burden of allergic rhinitis amongst UK patients 75% reported some impact of their allergic rhinitis symptoms on health-related quality of life. Allergic rhinitis currently affects 10-30% of the world population with prevalence and impact continuing to increase. This leads to substantial economic costs both of prescription medication and time taken off work by both patients and carers due to the disease. In view of this, there may be a substantial need for improved therapy or management to ensure that patients with allergic rhinitis can carry out a normal lifestyle.

The proposed study will evaluate the unmet therapy need in seasonal rhinitis by examining the current medication requirements of patients who suffer from seasonal grass-pollen hay fever and determining whether current therapies are sufficient for managing rhinitis.

This study aims to evaluate the unmet therapy need in seasonal rhinitis by -

1. Examining and describing current medication requirements
2. Quantifying the extent of co-prescribing of multiple agents
3. Comparing the effectiveness of current prescription drugs for managing and controlling patient's seasonal rhinitis and using changes in treatment during the hay fever season to determine the effectiveness of current therapy options.

for managing and controlling seasonal rhinitis in primary care patients who suffer from seasonal grass-pollen hay fever.

ELIGIBILITY:
Inclusion Criteria

The analysis will include patients who, at the index date, receive a therapy prescription for allergic rhinitis and have been diagnosed with a hay fever read code during their time at the practice. The following patients will be included within the study population:

(i)Patients receiving therapy: defined as those with a prescription for the increase or initiation of hay fever therapy during the hay fever season

(ii)Hay-fever code recorded ever

Exclusion criteria

(i)Patients taking maintenance oral steroids during the baseline period

(ii)Patients who only received LTRA during the study period and had already been receiving LTRA previously

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients will have seasonal rhinitis: defined as hay fever/rhinitis diagnosis during the hay fever season period and will be receiving therapy during the hay fever season
Sampling Method: Non-Probability Sample
Enrollment: 21203 (Actual)
Dates: Start 2013-01; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Co-prescribing | 31.11.12
  The proportion of patients managed at the index prescription date with more than one class of therapy
Treatment Outcomes | 10.12.12
  For those patients who receive a prescription for a diagnosis of seasonal rhinitis/ hay fever. The following outcomes will be measured -
  * Patients who remain on the same therapy
  * Patients who change therapy within same therapy group
  * Patients who add additional therapy from another therapy group
Number of Consultations | 10.12.12
  Defined as a consultation where an allergic rhinitis read code or hay fever code is recorded during the hay fever season.
Asthma Patients - Exacerbations: Clinical | 10.12.12
  where exacerbation is defined as an occurrence of the following:
  a)Lower respiratory related : Hospital attendance/admission OR A & E attendance; OR Out-of-hours attendance;
  * GP consultations for lower respiratory related tract infections;
  * Acute use of oral steroids .
Asthma Patients - Exacerbations: Severe | 10.12.12
  b)Asthma related -
  Hospital attendance/admission OR A & E attendance; OR Out-of-hours attendance; GP consultations for asthma related tract infections; Acute use of oral steroids
Costing Analysis | 15.01.13
  Descriptive analysis of costs at the first prescription and final prescription of the season. Comparing those who remain on same therapy and those who add therapy during the season.

CONTACTS AND LOCATIONS:
Overall Officials: David Price, Prof, MD, Principal Investigator — University of Aberdeen
Locations (1):
- Research in Real Life Ltd, Cambridge, United Kingdom

REFERENCES:
- [Background] Gupta R, Sheikh A, Strachan DP, Anderson HR. Burden of allergic disease in the UK: secondary analyses of national databases. Clin Exp Allergy. 2004 Apr;34(4):520-6. doi: 10.1111/j.1365-2222.2004.1935.x. PMID 15080802
- [Result] Van Cauwenberge P, Van Hoecke H, Kardos P, Price D, Waserman S. The current burden of allergic rhinitis amongst primary care practitioners and its impact on patient management. Prim Care Respir J. 2009 Mar;18(1):27-33. doi: 10.3132/pcrj.2008.00042. PMID 18622524
- [Result] Meltzer EO, Bukstein DA. The economic impact of allergic rhinitis and current guidelines for treatment. Ann Allergy Asthma Immunol. 2011 Feb;106(2 Suppl):S12-6. doi: 10.1016/j.anai.2010.10.014. PMID 21277528